CLINICAL TRIAL: NCT05172739
Title: Effect of a Perioperative Opioid Free Anaesthesia-Analgesia (OFA-A) Strategy on Surgical Stress Response and Immunomodulation in Elective VATS Lobectomy for NSCLC Lung Cancer: A Prospective Randomized Study
Brief Title: Opioid Free Anaesthesia-Analgesia Strategy on Surgical Stress and Immunomodulation in Elective VATS-Lobectomy for NSCLC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Crete (Other)
Responsible Party: Principal Investigator, Periklis Vasilos, Principal Investigator, University of Crete
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: OFA-Thoracic
Record Dates: First submitted 2021-11-13; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Systemic Inflammatory Response Syndrome; Postoperative Pain, Acute; Postoperative Pain, Chronic; Infections Postoperative; Opioid Use; Anesthesia; Non-small Cell Lung Cancer
Keywords: Opioid-free Anesthesia-Analgesia; Opioid-based Anesthesia-Analgesia; Cytokines; NSCLC; Hemodynamic stability; Immunomodulation; Inflammatory markers; Acute postoperative pain; Chronic postoperative pain
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Pain, Postoperative; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Administration of a multimodal anaesthetic opioid-free strategy that includes pregabalin, ketamine, dexmedetomidine, lidocaine, dexamethasone, magnesium sulphate, paracetamol and dexketoprofen is expected to affect the inflammatory and stress response, measured by levels of inflammatory markers and haemodynamic stability, when compared to conventional opioid based techniques. An Opioid-Free Anaesthesia-Analgesia strategy, is expected to also lead to an attenuated immunosuppression, due to the avoidance of opioids, whose administration has been corelated with immunosuppressive effects. An overall decreased inflammatory and stress response as expressed by reduced levels of inflammatory biomarkers and hemodynamic stability, is expected to decrease peripheral and central sensitization, contributing to better postoperative analgesia.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid-Based Anaesthesia Analgesia (Active Comparator): Premedication: IM Midazolam 0.05-0.07mg/kg. Anesthesia induction: Midazolam 0.03mg/kg, Propofol 2-3mg/kg, Fentanyl 1-2mcg/kg and Cisatracurium 0.2mg/kg or alternatively Rocuronium 0.6-1.2mg/ kg. Anesthesia maintenance: Desflurane set at approximately 1 MAC, Morphine 0.1-0.12mg/kg, Fentanyl 1-2mcg/kg during induction and 50-100mcg prn, Paracetamol 1g +/- Dexketoprofen trometamol 50mg, along with Ondansetron 4mg or Droperidol 0.625mg. Wound infiltration: Ropivacaine 75-150mg. Surgical ward: PCA pump with Morphine for the first 3 postoperative days. Additional postoperative analgesia: Paracetamol 1g 1x3 +/- Dexketoprofen trometamol 50mg 1x2. Rescue therapy only: Tramadol 50-100mg.
  Interventions: Drug: Opioid-Based Anesthesia-Analgesia Strategy
- Opioid-Free Anesthesia Analgesia (Active Comparator): Premedication: Pregabalin 150mg 1x2, IM Midazolam 0.05-0.07mg/kg. Anesthesia induction: Midazolam 0.03mg/kg, Dexmedetomidine 0.5-1mcg/kg, Lidocaine 1mg/kg, Propofol 2-3mg/kg, Ketamine 1-1.5mg/kg, Hyoscine 10mg, Cisatracurium 0.2mg/ kg or alternatively Rocuronium 0.6-1.2mg/kg, Magnesium sulphate 2.5-5g and Dexamethasone 8-16mg. Anesthesia maintenance: Desflurane set at ~1 MAC, Dexmedetomidine 0.5-1.2mcg/kg/h, Lidocaine 0.5-1mg/kg/h, Ketamine 0.3-0.5mg/kg prn, Paracetamol 1g +/- Dexketoprofen trometamol 50mg, and Ondansetron 4mg or Droperidol 0.625mg. Wound infiltration: Ropivacaine 75-150mg. Surgical ward: PCA pump with Ketamine, Lidocaine, Clonidine, Droperidol and Midazolam for the first 3 postoperative days. Additionally, Pregabalin 50mg per os 1x1 and 25mg 1x1, Paracetamol 1g 1x3 +/- Dexketoprofen trometamol 50mg 1x2. Rescue therapy only: Tramadol 50-100mg.
  Interventions: Drug: Opioid-free Anesthesia-Analgesia Strategy

INTERVENTIONS:
Drug: Opioid-Based Anesthesia-Analgesia Strategy — A perioperative Opioid-Based multimodal Anesthesia- Analgesia strategy will be implemented that incorporates the following pharmacological agents:
  Premedication: Midazolam, Anaesthesia induction & maintenance: Midazolam, Propofol, Fentanyl, Cisatracurium or alternatively Rocuronium, Desflurane, Morphine, Paracetamol, Dexketoprofen trometamol, Ondansetron or Droperidol, Ropivacaine Surgical ward: Morphine, Paracetamol, Dexketoprofen trometamol Rescue therapy only: Tramadol
  Other Names: Opioid-Based Anesthesia; OBA-A
  Arms: Opioid-Based Anaesthesia Analgesia
Drug: Opioid-free Anesthesia-Analgesia Strategy — A perioperative Opioid-Based multimodal Anesthesia- Analgesia strategy will be implemented that incorporates the following pharmacological agents:
  Premedication: Pregabalin, Midazolam, Anesthesia induction & maintenance: Midazolam, Dexmedetomidine, Lidocaine, Propofol, Ketamine, Hyoscine, Cisatracurium or alternatively Rocuronium, Magnesium sulphate, Dexamethasone, Desflurane, Paracetamol, Dexketoprofen trometamol, Ondansetron or Droperidol, Ropivacaine, Surgical ward: Ketamine, Lidocaine, Clonidine, Droperidol and Midazolam, Pregabalin, Paracetamol, Dexketoprofen trometamol Rescue therapy only: Tramadol
  Other Names: Opioid-Free Anesthesia; OFA-A
  Arms: Opioid-Free Anesthesia Analgesia

SUMMARY:
Lobectomy is a major, high-risk surgical procedure that in addition to one-lung ventilation (OLV) exerts a potent surgical stress response. An overwhelming immune cell recruitment may lead to excessive tissue damage, peripheral organ injury and immunoparesis. The effect of anesthesia on the immune system is modest, compared to the effects induced by major surgery. However, to an immunocompromised patient, due to cancer and/or other comorbidities, the immunosuppressive effects of anesthesia may increase the incidence of post-operative infections, morbidity, and mortality. Exogenous opioids have been correlated with immunosuppression, opioid-induced hyperalgesia, and respiratory depression, with deleterious outcomes. An Opioid-Free Anaesthesia-Analgesia (OFA-A) strategy is based on the administration of a variety of anaesthetic/analgesic and other pharmacological agents with different mechanisms of action, including immunomodulating and anti-inflammatory effects. Our basic hypothesis is that the implementation of a perioperative multimodal OFA-A strategy, will lead to an attenuated surgical stress response and attenuated immunosuppression, compared to a conventional Opioid-Based Anaesthesia-Analgesia (OBA-A) strategy. The aforementioned effects, are presumed to be associated with equal or improved analgesia and decreased incidence of postoperative infections compared to a perioperative OBA-A technique.

DETAILED DESCRIPTION:
Surgical manipulation and one lung ventilation (OLV) exert different and synergic effects to generate an inflammatory response during lung resection surgery. Surgery, such as lobectomies, often leads to severe immunosuppression that in turn can lead to infectious complications and sepsis. Both anesthesia-related and surgery-related perioperative measures may modulate the patient's immune response and lead to the activation of different components of the immune system. Anesthesia-induced activation, in particular of the adaptive immune system, may also induce persistent, postoperative immunosuppression. An overwhelming immune cell recruitment may lead to excessive tissue damage, peripheral organ injury and immunoparesis.

Opioid analgesia remains the corner stone of acute pain management in perioperative analgesic regimes. Opioid receptors are not only expressed in the central nervous system to regulate pain perception but also occur on immune and tumour cells. Exogenous opioid administration has been correlated with immunosuppression, opioid-induced hyperalgesia, and respiratory depression, with deleterious outcomes.

An Opioid-Free Anaesthesia-Analgesia (OFA-A) strategy is based on the administration of a variety of anaesthetic/analgesic and other pharmacological agents with different mechanisms of action, including immunomodulating and anti-inflammatory effects where at least one factor causes inhibition of central sensitization and at least another factor inhibits the peripheral sensitization of the nervous system, as a response to painful surgical stimuli. This combination of factors has to have a synergistic or additive effect so that best analgesic effects can be achieved with the lowest possible dosage.

Our basic hypothesis is that a perioperative OFA-A strategy on cancer patients undergoing VATS lung surgery for tumour resection will be accompanied by abolished or attenuated immunosuppression. The additional potential clinical implication of a perioperative OFA-A strategy is the avoidance of the onco-proliferative side effects of both exogenous and endogenous opioids, released by cytokine-mediated immune cell activation. Inflammatory response inhibition is expected to reduce the possibility of acute and chronic post-operative pain developement, compared to a perioperative Opioid-Based Anaesthesia- Analgesia (OBA-A) technique. Additionally, the aforementioned inflammatory response inhibition is expected to lead to an overall reduction of overall postoperative pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective VATS lobectomy
* early stage NSCLC (up to T3N1M0)

Exclusion Criteria:

* Immunocompromised patients
* previous lung surgery
* preoperative corticosteroid or immunosuppressive drug use
* uncontrolled Diabetes Mellitus
* cardiac failure (NYHA 3 and 4)
* preoperative infection (CRP >5mg/ml, WBC >10x10^9/L)
* preoperative anemia (Hb<12g/dl)
* chronic inflammatory diseases
* inflammatory bowel disease

Group-specific exclusion criteria:

* OFA-Α: perioperative opioid administration, within the study period
* OBA-Α: perioperative dexmedetomidine or lidocaine infusion, ketamine, gabapentinoid or corticosteroid administration within the study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Neutrophil to Lymphocyte ratio (NLR) | Preoperatively
  Neutrophil to Lymphocyte ratio (NLR) is a prognostic index that predicts patients' overall survival. Higher NLR has been correlated with worse outcome.
Platelet to Lymphocyte ratio (PLR) | Preoperatively
  Platelet to Lymphocyte ratio (PLR) is a prognostic index that predicts patients' overall survival. Higher PLR has been correlated with worse outcome.
Lymphocyte to monocyte ratio (LMR) | Preoperatively
  Lymphocyte to monocyte ratio (LMR) is a prognostic index that predicts patients' overall survival. Lower LMR has been correlated with worse outcome.
Advanced Lung Cancer Inflammation Index (ALI) | Preoperatively
  Advanced Lung Cancer Inflammation Index (ALI) is a prognostic index that predicts patients' recurrence-free survival and overall survival. ALI is calculated as (BMI x Alb / NLR) where BMI = body mass index, Alb = serum albumin, NLR (neutrophil lymphocyte ratio, a marker of systemic inflammation). Higher ALI scores have been correlated with worse outcome.
Systemic Immune Inflammation Index (SII) | Preoperatively
  Systemic Immune Inflammation Index (SII) is a prognostic index that predicts patients' overall survival. SII is calculated as follows: SII = platelet count × neutrophil/lymphocyte count. Higher SII scores have been correlated with worse outcome.
Prognostic Nutritional Index (PNI) | Preoperatively
  Prognostic Nutritional Index (PNI) is a prognostic index that predicts patients' overall survival. PNI is calculated as follows: PNI = 10 × serum albumin value (g/dL) + 0.005 × total lymphocyte count (per mm3) in the peripheral blood. Higher PNI scores have been correlated with worse outcome.
Surgical Stress Response - IL-6 - preoperatively | Preoperatively (as a baseline)
  Inflammatory response and stress response as quantified by IL-6 serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - IL-6 - end of surgery | End of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by IL-6 serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - IL-6 - 24 hours after the end of surgery | 24 hours after the end of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by IL-6 serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - IL-8 - preoperatively | Preoperatively (as a baseline)
  Inflammatory response and stress response as quantified by IL-8 serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - IL-8 - end of surgery | End of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by IL-8 serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - IL-8 - 24 hours after the end of surgery | 24 hours after the end of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by IL-8 serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - IL-10 - preoperatively | Preoperatively (as a baseline)
  Inflammatory response and stress response as quantified by IL-10 serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - IL-10 - end of surgery | End of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by IL-10 serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - IL-10 - 24 hours after the end of surgery | 24 hours after the end of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by IL-10 serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - TNF-a - preoperatively | Preoperatively (as a baseline)
  Inflammatory response and stress response as quantified by TNF-a serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - TNF-a - end of surgery | End of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by TNF-a serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - TNF-a - 24 hours after the end of surgery | 24 hours after the end of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by TNF-a serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - CRP - preoperatively | Preoperatively (as a baseline)
  Inflammatory response and stress response as quantified by CRP serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - CRP - end of surgery | End of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by CRP serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - CRP - 24 hours after the end of surgery | 24 hours after the end of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by CRP serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - WBC - preoperatively | Preoperatively (as a baseline)
  Inflammatory response and stress response as quantified by WBC count. Blood sample collection will take place in both study groups
Surgical Stress Response - WBC - end of surgery | End of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by WBC count. Blood sample collection will take place in both study groups
Surgical Stress Response - WBC - 24 hours after the end of surgery | 24 hours after the end of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by WBC count. Blood sample collection will take place in both study groups
Surgical Stress Response - AVP - preoperatively | Preoperatively (as a baseline)
  Inflammatory response and stress response as quantified by AVP serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - AVP - end of surgery | End of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by AVP serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - AVP - 24 hours after the end of surgery | 24 hours after the end of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by AVP serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - cortisol - preoperatively | Preoperatively (as a baseline)
  Inflammatory response and stress response as quantified by cortisol serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - cortisol - end of surgery | End of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by cortisol serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - cortisol - 24 hours after the end of surgery | 24 hours after the end of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by cortisol serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - HIF-1α- preoperatively | Preoperatively (as a baseline)
  Inflammatory response and stress response as quantified by HIF-1α serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - HIF-1α - end of surgery | End of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by HIF-1α serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - HIF-1α - 24 hours after the end of surgery | 24 hours after the end of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by HIF-1α serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - VEGF- preoperatively | Preoperatively (as a baseline)
  Inflammatory response and stress response as quantified by VEGF serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - VEGF- end of surgery | End of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by VEGF serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - VEGF - 24 hours after the end of surgery | 24 hours after the end of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by VEGF serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - NF-κB - preoperatively | Preoperatively (as a baseline)
  Inflammatory response and stress response as quantified by NF-κB serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - NF-κB - end of surgery | End of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by NF-κB serum levels. Blood sample collection will take place in both study groups
Surgical Stress Response - NF-κB - 24 hours after the end of surgery | 24 hours after the end of surgery (end of placement of last suture/ surgical clip on patient)
  Inflammatory response and stress response as quantified by NF-κB serum levels. Blood sample collection will take place in both study groups
Haemodynamic Stability - Mean PR | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Pulse Rate - PR. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Mean PR will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Minimum PR | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Pulse Rate - PR. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Minimum PR will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Maximum PR | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Pulse Rate - PR. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Maximum PR will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Standard Deviation PR | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Pulse Rate - PR. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Standard Deviation PR will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - PR Change Induction | 1 minute after anesthesia induction, compared to 1 minute prior
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Pulse Rate change 1 minute after anesthesia induction, compared to 1 minute prior. Data will be collected from a pulse contour analysis monitor.
Haemodynamic Stability - PR Change Incision | 1 minute after surgical incision, compared to 1 minute prior
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Pulse Rate change 1 minute after surgical incision, compared to 1 minute prior. Data will be collected from a pulse contour analysis monitor.
Haemodynamic Stability - Mean SBP | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Systolic Blood Pressure - SBP. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Mean SBP will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Minimum SBP | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Systolic Blood Pressure - SBP. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Minimum SBP will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Maximum SBP | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Systolic Blood Pressure - SBP. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Maximum SBP will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Standard Deviation SBP | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Systolic Blood Pressure - SBP. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Standard Deviation SBP will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - SBP Change Induction | 1 minute after anesthesia induction, compared to 1 minute prior
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Systolic Blood Pressure change 1 minute after anesthesia induction, compared to 1 minute prior. Data will be collected from a pulse contour analysis monitor.
Haemodynamic Stability - SBP Change Incision | 1 minute after surgical incision, compared to 1 minute prior
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Systolic Blood Pressure change 1 minute after surgical incision, compared to 1 minute prior. Data will be collected from a pulse contour analysis monitor.
Haemodynamic Stability - Mean DBP | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Diastolic Blood Pressure - DBP. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Mean DBP will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Minimum DBP | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Diastolic Blood Pressure - DBP. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Minimum DBP will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Maximum DBP | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Diastolic Blood Pressure - DBP. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Maximum DBP will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Standard Deviation DBP | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Diastolic Blood Pressure - DBP. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Standard Deviation DBP will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - DBP change induction | 1 minute after anesthesia induction, compared to 1 minute prior
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Diastolic Blood Pressure change 1 minute after anesthesia induction, compared to 1 minute prior. Data will be collected from a pulse contour analysis monitor.
Haemodynamic Stability - DBP change incision | 1 minute after surgical incision, compared to 1 minute prior
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Diastolic Blood Pressure change 1 minute after surgical incision, compared to 1 minute prior. Data will be collected from a pulse contour analysis monitor.
Haemodynamic Stability - Mean MBP | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Mean Blood Pressure - MBP. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Mean MBP will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Minimum MBP | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Mean Blood Pressure - MBP. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Minimum MBP will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Maximum MBP | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Mean Blood Pressure - MBP. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Maximum MBP will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Standard Deviation MBP | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Mean Blood Pressure - MBP. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Standard Deviation MBP will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - MBP change induction | 1 minute after anesthesia induction, compared to 1 minute prior
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Mean Blood Pressure change 1 minute after anesthesia induction, compared to 1 minute prior. Data will be collected from a pulse contour analysis monitor.
Haemodynamic Stability - MBP change incision | 1 minute after surgical incision, compared to 1 minute prior
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Mean Blood Pressure change 1 minute after surgical incision, compared to 1 minute prior. Data will be collected from a pulse contour analysis monitor.
Haemodynamic Stability - Mean CO | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Cardiac Output - CO. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Mean CO will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Minimum CO | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Cardiac Output - CO. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Minimum CO will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Maximum CO | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Cardiac Output - CO. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Maximum CO will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Standard Deviation CO | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Cardiac Output - CO. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Standard Deviation CO will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Mean CI | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Cardiac Index - CI. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Mean CI will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Minimum CI | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Cardiac Index - CI. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Minimum CI will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Maximum CI | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Cardiac Index - CI. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Maximum CI will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Standard Deviation CI | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Cardiac Index - CI. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Standard Deviation CI will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Mean SV | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Stroke Volume - SV. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Mean SV will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Minimum SV | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Stroke Volume - SV. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Minimum SV will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Maximum SV | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Stroke Volume - SV. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Maximum SV will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Standard Deviation SV | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Stroke Volume - SV. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Standard Deviation SV will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Mean SVV | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Stroke Volume Variation - SVV. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Mean SVV will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Minimum SVV | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Stroke Volume Variation - SVV. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Minimum SVV will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Maximum SVV | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Stroke Volume Variation - SVV. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Maximum SVV will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Standard Deviation SVV | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Stroke Volume Variation - SVV. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Standard Deviation SVV will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Mean SVI | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Stroke Volume Index - SVI. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Mean SVI will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Minimum SVI | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Stroke Volume Index - SVI. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Minimum SVI will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Maximum SVI | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Stroke Volume Index - SVI. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Maximum SVI will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Standard Deviation SVI | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/ surgical clip on patient), assessed up to 8 hours]
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Stroke Volume Index - SVI. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Standard Deviation SVI will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Tachycardia | Intraoperatively, assessed up to 4 hours.
  Intraoperative Tachycardia (defined as PR≥ 100 bpm), with episodes lasting ≥1 minute. Data will be reported in total seconds of intraoperative tachycardia.
Haemodynamic Stability - Bradycardia | Intraoperatively, assessed up to 4 hours.
  Intraoperative Bradycardia (defined as PR≤ 60 bpm), with episodes lasting ≥1 minute. Data will be reported in total seconds of intraoperative bradycardia.
Haemodynamic Stability - Hypotension | Intraoperatively, assessed up to 6 hours.
  Intraoperative Hypotension (defined as SBP≤100mmHg or ≤70% of preoperative Baseline), with episodes lasting ≥1 minute. All patients will have a 5 minute preoperative SBP baseline, with measurements every 20 seconds. Intraoperative data will be compared to the mean preoperative 5 minute SPB baseline. Data will be reported in total seconds of intraoperative hypotension.
Haemodynamic Stability - Hypertension | Intraoperatively, assessed up to 6 hours.
  Intraoperative Hypertension (defined as SBP ≥130% of preoperative Baseline), with episodes lasting ≥1 minute. All patients will have a 5 minute preoperative SBP baseline, with measurements every 20 seconds. Intraoperative data will be compared to the mean preoperative 5 minute SPB baseline. Data will be reported in total seconds of intraoperative hypertension.
Haemodynamic Stability - Fluid requirements - Crystalloids - Intraoperatively | Intraoperatively, assessed up to 6 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Crystalloid Fluid Requirements.
Haemodynamic Stability - Fluid requirements - Colloids - Intraoperatively | Intraoperatively, assessed up to 6 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Colloid Fluid Requirements.
Haemodynamic Stability - Fluid requirements - Concentrated RBCs - Intraoperatively | Intraoperatively, assessed up to 6 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Concentrated Red Blood Cell unit Requirements.
Haemodynamic Stability - Fluid requirements - Plasma - Intraoperatively | Intraoperatively, assessed up to 6 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Plasma unit Requirements.
Haemodynamic Stability - Fluid requirements - Platelets - Intraoperatively | Intraoperatively, assessed up to 6 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Platelet unit Requirements.
Haemodynamic Stability - Blood Loss - Intraoperatively | Intraoperatively, assessed up to 6 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Blood Loss
Haemodynamic Stability - Fluid Balance - Intraoperatively | Intraoperatively, assessed up to 6 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Fluid Balance
Haemodynamic Stability - Vasoactive Requirements - Adrenaline - Intraoperatively | Intraoperatively, assessed up to 6 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Adrenaline requirements
Haemodynamic Stability - Vasoactive Requirements - Noradrenaline - Intraoperatively | Intraoperatively, assessed up to 6 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Noradrenaline requirements
Haemodynamic Stability - Vasoactive Requirements - Ephedrine - Intraoperatively | Intraoperatively, assessed up to 6 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Ephedrine requirements
Haemodynamic Stability - Vasoactive Requirements - Phenylephrine - Intraoperatively | Intraoperatively, assessed up to 6 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Phenylephrine requirements
Haemodynamic Stability - Vasoactive Requirements - Dopamine - Intraoperatively | Intraoperatively, assessed up to 6 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Dopamine requirements
Haemodynamic Stability - Vasoactive Requirements - Dobutamine - Intraoperatively | Intraoperatively, assessed up to 6 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Dobutamine requirements
Haemodynamic Stability - Vasoactive Requirements - Nitroglycerine - Intraoperatively | Intraoperatively, assessed up to 6 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Nitroglycerine requirements

SECONDARY OUTCOMES:
Acute postoperative pain - Numerical Rating Scale (NRS) - Immediately Postoperatively | Immediately postoperatively
  Evaluation of patients' pain using scales: Numerical Rating Scale (NRS). The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Acute postoperative pain - Numerical Rating Scale (NRS) - First postoperative day | First postoperative day
  Evaluation of patients' pain using scales: Numerical Rating Scale (NRS). The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Acute postoperative pain - Numerical Rating Scale (NRS) - Second postoperative day | Second postoperative day
  Evaluation of patients' pain using scales: Numerical Rating Scale (NRS). The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Acute postoperative pain - Numerical Rating Scale (NRS) - Third postoperative day | Third postoperative day
  Evaluation of patients' pain using scales: Numerical Rating Scale (NRS). The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Acute postoperative pain - Critical Care Pain Observation Tool (CPOT) - Immediately Postoperatively | Immediately postoperatively
  Evaluation of patients' pain using scales: Critical Care Pain Observation Tool (CPOT). The scale consists of four behavioral domains: facial expression, body movements, muscle tension and compliance with the ventilation for intubated patients or vocalization for extubated patients. Patient's behavior in each domain is scored between 0 and 2. The possible total score ranges from 0 (no pain) to 8 (maximum pain).
Acute postoperative pain - Critical Care Pain Observation Tool (CPOT) - First postoperative day | First postoperative day
  Evaluation of patients' pain using scales: Critical Care Pain Observation Tool (CPOT). The scale consists of four behavioral domains: facial expression, body movements, muscle tension and compliance with the ventilation for intubated patients or vocalization for extubated patients. Patient's behavior in each domain is scored between 0 and 2. The possible total score ranges from 0 (no pain) to 8 (maximum pain).
Acute postoperative pain - Critical Care Pain Observation Tool (CPOT) - Second postoperative day | Second postoperative day
  Evaluation of patients' pain using scales: Critical Care Pain Observation Tool (CPOT). The scale consists of four behavioral domains: facial expression, body movements, muscle tension and compliance with the ventilation for intubated patients or vocalization for extubated patients. Patient's behavior in each domain is scored between 0 and 2. The possible total score ranges from 0 (no pain) to 8 (maximum pain).
Acute postoperative pain - Critical Care Pain Observation Tool (CPOT) - Third postoperative day | Third postoperative day
  Evaluation of patients' pain using scales: Critical Care Pain Observation Tool (CPOT). The scale consists of four behavioral domains: facial expression, body movements, muscle tension and compliance with the ventilation for intubated patients or vocalization for extubated patients. Patient's behavior in each domain is scored between 0 and 2. The possible total score ranges from 0 (no pain) to 8 (maximum pain).
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Intolerable - First postoperative day | First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Intolerable" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Intolerable - Second postoperative day | Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Intolerable" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Intolerable - Third postoperative day | Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Intolerable" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Tolerable with discomfort - First postoperative day | First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Tolerable with Discomfort" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Tolerable with discomfort - Second postoperative day | Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Tolerable with Discomfort" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Tolerable with discomfort - Third postoperative day | Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Tolerable with Discomfort" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Comfortably manageable - First postoperative day | First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Comfortably manageable" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Comfortably manageable - Second postoperative day | Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Comfortably manageable" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Comfortably manageable - Third postoperative day | Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Comfortably manageable" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Negligible Pain - First postoperative day | First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Negligible Pain" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Negligible Pain - Second postoperative day | Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Negligible Pain" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Negligible Pain - Third postoperative day | Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Negligible Pain" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Change in Pain - Getting Worse - First postoperative day | First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to changes in pain perception by patients, available answers will be:
  1. Getting worse
  2. About the same
  3. Getting better
  The percentage of patients that report pain that is "Getting worse" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Change in Pain - Getting Worse - Second postoperative day | Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to changes in pain perception by patients, available answers will be:
  1. Getting worse
  2. About the same
  3. Getting better
  The percentage of patients that report pain that is "Getting worse" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Change in Pain - Getting Worse - Third postoperative day | Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to changes in pain perception by patients, available answers will be:
  1. Getting worse
  2. About the same
  3. Getting better
  The percentage of patients that report pain that is "Getting worse" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Change in Pain - About the same - First postoperative day | First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to changes in pain perception by patients, available answers will be:
  1. Getting worse
  2. About the same
  3. Getting better
  The percentage of patients that report pain that is "About the same" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Change in Pain - About the same - Second postoperative day | Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to changes in pain perception by patients, available answers will be:
  1. Getting worse
  2. About the same
  3. Getting better
  The percentage of patients that report pain that is "About the same" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Change in Pain - About the same - Third postoperative day | Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to changes in pain perception by patients, available answers will be:
  1. Getting worse
  2. About the same
  3. Getting better
  The percentage of patients that report pain that is "About the same" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Change in Pain - Getting better - First postoperative day | First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to changes in pain perception by patients, available answers will be:
  1. Getting worse
  2. About the same
  3. Getting better
  The percentage of patients that report pain that is "Getting Better" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Change in Pain - Getting better - Second postoperative day | Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to changes in pain perception by patients, available answers will be:
  1. Getting worse
  2. About the same
  3. Getting better
  The percentage of patients that report pain that is "Getting Better" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Change in Pain - Getting better - Third postoperative day | Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to changes in pain perception by patients, available answers will be:
  1. Getting worse
  2. About the same
  3. Getting better
  The percentage of patients that report pain that is "Getting Better" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Pain control - Inadequate pain control - First postoperative day | First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to pain control reported by patients, available answers will be:
  1. Inadequate pain control
  2. Effective, just about right
  3. Would like to reduce medication
  The percentage of patients that report "Inadequate pain control" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Pain control - Inadequate pain control - Second postoperative day | Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to pain control reported by patients, available answers will be:
  1. Inadequate pain control
  2. Effective, just about right
  3. Would like to reduce medication
  The percentage of patients that report "Inadequate pain control" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Pain control - Inadequate pain control - Third postoperative day | Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to pain control reported by patients, available answers will be:
  1. Inadequate pain control
  2. Effective, just about right
  3. Would like to reduce medication
  The percentage of patients that report "Inadequate pain control" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Pain control - Effective, just about right - First postoperative day | First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to pain control reported by patients, available answers will be:
  1. Inadequate pain control
  2. Effective, just about right
  3. Would like to reduce medication
  The percentage of patients that report "Effective, just about right" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Pain control - Effective, just about right - Second postoperative day | Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to pain control reported by patients, available answers will be:
  1. Inadequate pain control
  2. Effective, just about right
  3. Would like to reduce medication
  The percentage of patients that report "Effective, just about right" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Pain control - Effective, just about right - Third postoperative day | Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to pain control reported by patients, available answers will be:
  1. Inadequate pain control
  2. Effective, just about right
  3. Would like to reduce medication
  The percentage of patients that report "Effective, just about right" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Pain control - Would like to reduce medication - First postoperative day | First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to pain control reported by patients, available answers will be:
  1. Inadequate pain control
  2. Effective, just about right
  3. Would like to reduce medication
  The percentage of patients that report "Would like to reduce medication" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Pain control - Would like to reduce medication - Second postoperative day | Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to pain control reported by patients, available answers will be:
  1. Inadequate pain control
  2. Effective, just about right
  3. Would like to reduce medication
  The percentage of patients that report "Would like to reduce medication" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Pain control - Would like to reduce medication - Third postoperative day | Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to pain control reported by patients, available answers will be:
  1. Inadequate pain control
  2. Effective, just about right
  3. Would like to reduce medication
  The percentage of patients that report "Would like to reduce medication" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Can't do anything because of pain - First postoperative day | First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Can't do anything because of pain" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Can't do anything because of pain - Second postoperative day | Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Can't do anything because of pain" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Can't do anything because of pain - Third postoperative day | Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Can't do anything because of pain" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Pain keeps me from doing most of what I need to do - First postoperative day | First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Pain keeps me from doing most of what I need to do" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Pain keeps me from doing most of what I need to do - Second postoperative day | Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Pain keeps me from doing most of what I need to do" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Pain keeps me from doing most of what I need to do - Third postoperative day | Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Pain keeps me from doing most of what I need to do" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Can do most things, but pain gets in the way of some - First postoperative day | First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Can do most things, but pain gets in the way of some" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Can do most things, but pain gets in the way of some - Second postoperative day | Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Can do most things, but pain gets in the way of some" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Can do most things, but pain gets in the way of some - Third postoperative day | Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Can do most things, but pain gets in the way of some" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Can do everything I need to do - First postoperative day | First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Can do everything I need to do" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Can do everything I need to do - Second postoperative day | Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Can do everything I need to do" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Can do everything I need to do - Third postoperative day | Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Can do everything I need to do" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Sleep - Awake with pain most of the night - First postoperative day | First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to sleep, if the pain is waking patients up, available answers will be:
  1. Awake with pain most of the night
  2. Awake with occasional pain
  3. Normal sleep
  The percentage of patients whose sleep is reported as "Awake with pain most of the night" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Sleep - Awake with pain most of the night - Second postoperative day | Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to sleep, if the pain is waking patients up, available answers will be:
  1. Awake with pain most of the night
  2. Awake with occasional pain
  3. Normal sleep
  The percentage of patients whose sleep is reported as "Awake with pain most of the night" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Sleep - Awake with pain most of the night - Third postoperative day | Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to sleep, if the pain is waking patients up, available answers will be:
  1. Awake with pain most of the night
  2. Awake with occasional pain
  3. Normal sleep
  The percentage of patients whose sleep is reported as "Awake with pain most of the night" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Sleep - Awake with occasional pain - First postoperative day | First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to sleep, if the pain is waking patients up, available answers will be:
  1. Awake with pain most of the night
  2. Awake with occasional pain
  3. Normal sleep
  The percentage of patients whose sleep is reported as " Awake with occasional pain" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Sleep - Awake with occasional pain - Second postoperative day | Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to sleep, if the pain is waking patients up, available answers will be:
  1. Awake with pain most of the night
  2. Awake with occasional pain
  3. Normal sleep
  The percentage of patients whose sleep is reported as " Awake with occasional pain" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Sleep - Awake with occasional pain - Third postoperative day | Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to sleep, if the pain is waking patients up, available answers will be:
  1. Awake with pain most of the night
  2. Awake with occasional pain
  3. Normal sleep
  The percentage of patients whose sleep is reported as " Awake with occasional pain" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Sleep - Normal sleep - First postoperative day | First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to sleep, if the pain is waking patients up, available answers will be:
  1. Awake with pain most of the night
  2. Awake with occasional pain
  3. Normal sleep
  The percentage of patients whose sleep is reported as "Normal sleep" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Sleep - Normal sleep - Second postoperative day | Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to sleep, if the pain is waking patients up, available answers will be:
  1. Awake with pain most of the night
  2. Awake with occasional pain
  3. Normal sleep
  The percentage of patients whose sleep is reported as "Normal sleep" will be reported
Acute postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Sleep - Normal sleep - Third postoperative day | Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to sleep, if the pain is waking patients up, available answers will be:
  1. Awake with pain most of the night
  2. Awake with occasional pain
  3. Normal sleep
  The percentage of patients whose sleep is reported as "Normal sleep" will be reported
Analgesic Requirements - First postoperative day | First postoperative day
  Evaluation of patients' pain by recording the number of times that rescue analgesia (tramadol) was required.
Analgesic Requirements - Second postoperative day | Second postoperative day
  Evaluation of patients' pain by recording the number of times that rescue analgesia (tramadol) was required.
Analgesic Requirements - Third postoperative day | Third postoperative day
  Evaluation of patients' pain by recording the number of times that rescue analgesia (tramadol) was required.
Postoperative Pulmonary Complications - Aspiration Pneumonitis | From the first postoperative day, until the fifth postoperative day
  Aspiration pneumonitis (defined as respiratory failure after the inhalation of regurgitated gastric contents)
Postoperative Pulmonary Complications - Moderate respiratory failure | From the first postoperative day, until the fifth postoperative day
  Moderate respiratory failure (SpO2 < 90% or PaO2 < 60 mmHg for 10 min in room air, responding to oxygen > 2 L/min)
Postoperative Pulmonary Complications - Severe respiratory failure | From the first postoperative day, until the fifth postoperative day
  Severe respiratory failure (need for non-invasive or invasive mechanical ventilation due to poor oxygenation)
Postoperative Pulmonary Complications - ARDS | From the first postoperative day, until the fifth postoperative day
  Adult respiratory distress syndrome (mild, moderate, or severe according to the Berlin definition)
Postoperative Pulmonary Complications - Pulmonary Infection | From the first postoperative day, until the fifth postoperative day
  Pulmonary infection (defined as new or progressive radiographic infiltrate plus at least two of the following: antibiotic treatment, tympanic temperature > 38 °C, leukocytosis or leucopenia (white blood cell (WBC) count < 4000 cells/mm3 or > 12,000 cells/mm3) and/or purulent secretions)
Postoperative Pulmonary Complications - Atelectasis | From the first postoperative day, until the fifth postoperative day
  Atelectasis (suggested by lung opacification with shift of the mediastinum, hilum, or hemidiaphragm towards the affected area, and compensatory over-inflation in the adjacent non-atelectatic lung)
Postoperative Pulmonary Complications - Cardiopulmonary edema | From the first postoperative day, until the fifth postoperative day
  Cardiopulmonary edema (defined as clinical signs of congestion, including dyspnea, edema, rales, and jugular venous distention, with the chest x-ray demonstrating increase in vascular markings and diffuse alveolar interstitial infiltrates)
Postoperative Pulmonary Complications - Pleural effusion | From the first postoperative day, until the fifth postoperative day
  Pleural effusion (chest x-ray demonstrating blunting of the costophrenic angle, loss of the sharp silhouette of the ipsilateral hemidiaphragm in upright position, evidence of displacement of adjacent anatomical structures, or (in supine position) a hazy opacity in one hemithorax with preserved vascular shadows)
Postoperative Pulmonary Complications - Pneumothorax | From the first postoperative day, until the fifth postoperative day
  Pneumothorax (defined as air in the pleural space with no vascular bed surrounding the visceral pleura)
Postoperative Pulmonary Complications - Pulmonary Infiltrates | From the first postoperative day, until the fifth postoperative day
  Pulmonary infiltrates (chest x-ray demonstrating new monolateral or bilateral infiltrate without other clinical signs)
Postoperative Pulmonary Complications - Prolonged air leakage | From the first postoperative day, until the fifth postoperative day
  Prolonged air leakage (air leak requiring at least 7 days of postoperative chest tube drainage)
Postoperative Pulmonary Complications - Purulent pleuritic | From the first postoperative day, until the fifth postoperative day
  Purulent pleuritic (receiving antibiotics for a suspected infection, as far as not explained by the preoperative patient condition alone)
Postoperative Pulmonary Complications - Pulmonary embolism | From the first postoperative day, until the fifth postoperative day
  Pulmonary embolism (as documented by pulmonary arteriogram or autopsy, or supported by ventilation/perfusion radioisotope scans, or documented by echocardiography and receiving specific therapy)
Postoperative Pulmonary Complications - Lung hemorrhage | From the first postoperative day, until the fifth postoperative day
  Lung hemorrhage (bleeding through the chest tubes requiring reoperation, or three or more red blood cell packs)
Chronic postoperative pain - Pain Detect | Three months after the end of surgery
  Evaluation of patients' pain using the standardized "Pain Detect" questionnaire. The "Pain Detect" questionnaire has been standardized for screening the presence of a neuropathic pain component. Patients will be interviewed by phone interview, 3 months after the end of surgery. The possible score a patient can have, ranges from 0 to 38.

CONTACTS AND LOCATIONS:
Overall Officials: Vasileia Nyktari, MD, PhD, Study Chair — University of Crete, Medical school
Locations (1):
- University of Crete, Heraklion, Crete, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanchez-Pedrosa G, Vara Ameigeiras E, Casanova Barea J, Rancan L, Simon Adiego CM, Garutti Martinez I. Role of surgical manipulation in lung inflammatory response in a model of lung resection surgery. Interact Cardiovasc Thorac Surg. 2018 Dec 1;27(6):870-877. doi: 10.1093/icvts/ivy198. PMID 29945217
- [Background] Schneemilch CE, Hachenberg T, Ansorge S, Ittenson A, Bank U. Effects of different anaesthetic agents on immune cell function in vitro. Eur J Anaesthesiol. 2005 Aug;22(8):616-23. doi: 10.1017/s0265021505001031. PMID 16119599
- [Background] Homburger JA, Meiler SE. Anesthesia drugs, immunity, and long-term outcome. Curr Opin Anaesthesiol. 2006 Aug;19(4):423-8. doi: 10.1097/01.aco.0000236143.61593.14. PMID 16829725
- [Background] Kurosawa S, Kato M. Anesthetics, immune cells, and immune responses. J Anesth. 2008;22(3):263-77. doi: 10.1007/s00540-008-0626-2. Epub 2008 Aug 7. PMID 18685933
- [Background] Calogero AE, Norton JA, Sheppard BC, Listwak SJ, Cromack DT, Wall R, Jensen RT, Chrousos GP. Pulsatile activation of the hypothalamic-pituitary-adrenal axis during major surgery. Metabolism. 1992 Aug;41(8):839-45. doi: 10.1016/0026-0495(92)90164-6. PMID 1640860
- [Background] Ninkovic J, Roy S. Role of the mu-opioid receptor in opioid modulation of immune function. Amino Acids. 2013 Jul;45(1):9-24. doi: 10.1007/s00726-011-1163-0. Epub 2011 Dec 15. PMID 22170499
- [Background] Kosciuczuk U, Knapp P, Lotowska-Cwiklewska AM. Opioid-induced immunosuppression and carcinogenesis promotion theories create the newest trend in acute and chronic pain pharmacotherapy. Clinics (Sao Paulo). 2020 Mar 23;75:e1554. doi: 10.6061/clinics/2020/e1554. eCollection 2020. PMID 32215455
- [Background] Plein LM, Rittner HL. Opioids and the immune system - friend or foe. Br J Pharmacol. 2018 Jul;175(14):2717-2725. doi: 10.1111/bph.13750. Epub 2017 Mar 23. PMID 28213891
- [Background] Vallejo R, de Leon-Casasola O, Benyamin R. Opioid therapy and immunosuppression: a review. Am J Ther. 2004 Sep-Oct;11(5):354-65. doi: 10.1097/01.mjt.0000132250.95650.85. PMID 15356431
- [Background] Finley MJ, Happel CM, Kaminsky DE, Rogers TJ. Opioid and nociceptin receptors regulate cytokine and cytokine receptor expression. Cell Immunol. 2008 Mar-Apr;252(1-2):146-54. doi: 10.1016/j.cellimm.2007.09.008. Epub 2008 Feb 14. PMID 18279847
- [Background] Parkhill AL, Bidlack JM. Reduction of lipopolysaccharide-induced interleukin-6 production by the kappa opioid U50,488 in a mouse monocyte-like cell line. Int Immunopharmacol. 2006 Jun;6(6):1013-9. doi: 10.1016/j.intimp.2006.01.012. Epub 2006 Feb 17. PMID 16644488
- [Background] Busch-Dienstfertig M, Stein C. Opioid receptors and opioid peptide-producing leukocytes in inflammatory pain--basic and therapeutic aspects. Brain Behav Immun. 2010 Jul;24(5):683-94. doi: 10.1016/j.bbi.2009.10.013. Epub 2009 Oct 29. PMID 19879349
- [Background] Stein C, Kuchler S. Non-analgesic effects of opioids: peripheral opioid effects on inflammation and wound healing. Curr Pharm Des. 2012;18(37):6053-69. doi: 10.2174/138161212803582513. PMID 22747536